CLINICAL TRIAL: NCT02558439
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging 24-Week Study to Evaluate the Safety and Efficacy of a Single Injection of CNTX-4975 in Subjects With Chronic, Moderate to Severe Osteoarthritis Knee Pain
Brief Title: Study to Evaluate the Safety and Efficacy of CNTX-4975 in Subjects With Chronic, Moderate to Severe Osteoarthritis Knee Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centrexion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4975-OA-502
Record Dates: First submitted 2015-09-20; First posted 2015-09-24 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — CNTX-4975

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Placebo (Placebo Comparator): Subjects will receive a single injection of placebo into the index knee following local anesthesia and adjunct joint cooling.
  Interventions: Other: Placebo
- 0.5 mg CNTX-4975 (Experimental): Subjects will receive a single injection of 0.5 mg CNTX-4975 into the index knee following local anesthesia and adjunct joint cooling.
  Interventions: Drug: CNTX-4975
- 1.0 mg CNTX-4975 (Experimental): Subjects will receive a single injection of 1.0 mg CNTX-4975 into the index knee following local anesthesia and adjunct joint cooling.
  Interventions: Drug: CNTX-4975

INTERVENTIONS:
Drug: CNTX-4975
  Arms: 0.5 mg CNTX-4975; 1.0 mg CNTX-4975
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a single injection of CNTX-4975 in subjects with chronic, moderate to severe osteoarthritis knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Radiography of both knees with a posterior-anterior, fixed flexion view taken during the Screening period. The index knee must show evidence of chronic OA.
* Moderate to severe pain in the index knee associated with OA must be stable for a minimum of 2 months prior to Screening, as assessed by the Investigator.
* A specified mean pain score in the index knee over the 7 days prior to dosing, based on question A1 of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC A1).
* Specified baseline and screening scores on the WOMAC A1
* Body Mass Index ≤ 45 kg/m2.
* Subjects must have had a therapeutic failure (no relief, or inadequate relief), and/or AEs resulting in stopping treatment, and/or contraindication to the standard of care appropriate to the severity of the index knee OA pain they are experiencing.

Exclusion Criteria:

* Joint replacement surgery of the index knee at any time, or open surgery of the index knee in the past 12 months.
* Prior arthroscopic surgery of the index knee within 3 months of Screening.
* Any painful conditions of the index knee due to joint disease other than OA.
* Mild pain in the non-index knee when walking.
* Other chronic pain anywhere in the body that requires the use of analgesic medications.
* Secondary OA of the index knee due to acute traumatic injury.
* Significant current or past instability (e.g., cruciate ligament tear or rupture or previous repair) or misalignment (> 10 degrees varus or valgus) of the index knee
* Has used topical capsaicin on the index knee within 90 days of Screening.
* Corticosteroid injection in the index knee within 90 days of Screening.
* Received IA viscosupplementation (e.g., Synvisc®, Hyalgan®) within 90 days of Screening.
* Prior participation in an ALGRX 4975 or CNTX-4975 study.
* Has any of the following characteristics:

  1. active or historic substance use disorder within the previous year as defined by the Diagnostic and Statistical Manual for Mental Health Disorders, fifth edition, or
  2. tests positive upon urine drug screen for a substance of abuse.
* Has moderate to severe depression or anxiety.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline through Week 12 in average knee index pain with walking over previous 24 hours using WOMAC A1 question in subjects treated with CNTX-4975 1.0 mg compared to placebo in subjects with osteoarthritis (OA) of the knee | At 12 Weeks

SECONDARY OUTCOMES:
Change from Baseline through Week 12 in average index knee pain with walking using WOMAC A1 question in subjects treated with CNTX 0.5 mg compared to placebo | At 12 Weeks
Change from Baseline to each study visit through Week 24 in average index knee pain with walking using WOMAC A1 in subjects treated with CNTX-4975 compared to placebo | Up to 24 weeks
Change from Baseline through Week 4 in the average index knee pain with walking using the WOMAC A1 question | Up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Advanced Arizona Clinical Research, Tucson, Arizona
  - Dream Team Clinical Research, LLC, Anaheim, California
  - Hope Clinical Research, LLC, Canoga Park, California
  - TriWest Research Associates, El Cajon, California
  - BioSolutions Clinical Research Center, La Mesa, California
  - Axis Clinical Trials, Los Angeles, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Finlay Research Clinic, Hialeah, Florida
  - Eastern Research, Hialeah, Florida
  - Sunrise Medical Research, Lauderdale Lakes, Florida
  - M&M Medical Center, Inc, Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - Compass Research, LLC, The Villages, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Drug Trials America, Hartsdale, New York
  - Manhattan Medical Research Practice, New York, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - University Orthopedics Center, Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania

REFERENCES:
- [Derived] Stevens RM, Ervin J, Nezzer J, Nieves Y, Guedes K, Burges R, Hanson PD, Campbell JN. Randomized, Double-Blind, Placebo-Controlled Trial of Intraarticular Trans-Capsaicin for Pain Associated With Osteoarthritis of the Knee. Arthritis Rheumatol. 2019 Sep;71(9):1524-1533. doi: 10.1002/art.40894. Epub 2019 Jul 17. PMID 30888737